CLINICAL TRIAL: NCT04479449
Title: A Prospective, Randomized, Double-blind Phase 2b Clinical Trial to Investigate the Efficacy and Safety of SP-8203 in Patients With Acute Ischemic Stroke Requiring Recombinant Tissue Plasminogen Activator (rtPA) Standard of Care
Brief Title: Efficacy and Safety of SP-8203 in Patients With Ischemic Stroke Requiring rtPA
Acronym: SP-8203-2002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-8203-2002
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke
Keywords: SP-8203 (Otaplimastat); rtPA (recombinant tissue Plasminogen Activator)
MeSH Terms: conditions — Ischemic Stroke | interventions — otaplimastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-8203 (Experimental): SP-8203 80 mg (40 mg/dose twice a day for three days)
  Interventions: Drug: SP-8203
- Placebo (Placebo Comparator): Placebo group: twice a day for three days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-8203 — SP-8203 80 mg will be intravenously administered as 40 mg/dose twice daily (intervals of 12 hours)
  Other Names: Otaplimastat (SP-8203)
  Arms: SP-8203
Drug: Placebo — Placebo will be intravenously administered twice daily (intervals of 12 hours)
  Arms: Placebo

SUMMARY:
This clinical trial is designed to evaluate the efficacy and safety of the combination therapy of SP-8203 (Otaplimastat) and recombinant tissue Plasminogen Activator (rtPA) standard of care. In this clinical trial, rtPA will be injected intravenously using an infusion device. If reperfusion is not occur in spite of rtPA therapy, endovascular therapy can be performed.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate the efficacy and safety of the combination therapy of SP-8203 and rtPA in patients with acute ischemic stroke receiving rtPA standard of care.

As the standard procedure of rtPA therapy, rtPA will be injected intravenously using an infusion device. When reperfusion is not achieved in spite of rtPA therapy, endovascular therapy can be performed according to the judgment of a site investigator.

A total of 178 subjects will be enrolled in double-blind, randomized and parallel design with 89 subjects assigned to 80 mg/day SP-8203 group or placebo group, respectively.

If a subject, who is able to be enrolled, has neurologic deficit of ≥4 point on the National Institute of Health Stroke Scale (NIHSS) score and give his/her consent to participate in the trial, each treatment is administered after the investigational product is randomly assigned by institution after sequential allocation. The randomization number of patients is the same as the assigned number of the investigational product administered to the patients. The subject will receive the Investigational products a total of 6 times, with 12 hours intervals. Only for the patients who consent, blood sample will be taken after the sixth administration of the Investigational product for pharmacokinetic and pharmacodynamics analysis. For pharmacokinetic profile analysis, blood sample will be taken at 0~5, 30±5, and 120±5 minutes after the complete sixth administration of the investigational products. For pharmacodynamic profile analysis, blood sample will be taken at between 24 to 48 hours after the first administration, at 0 minute after the sixth administration and at 4th week visit. The first blood sampling time is set to after 24 hours because of the patient's stability, but it can be performed before the investigational product has been administered in accordance with the judgment of the investigators.

The subject will have brain initial Magnetic Resonance Imaging (MRI) and Magnetic Resonance Angiography (MRA) performed within 6 hours before and after the administration of investigational product, and brain Computed Tomography (CT) will be performed at 24±3 hours after completion of the first administration of investigational products.

Brain MRI and MRA will be followed-up on Day 5, and additionally the subject will make a visit for close monitoring for his/her neurologic condition at 4th week and 12th week. Thereafter, all the procedures of the clinical trial will be completed.

When unexpected serious adverse reaction occurs during the clinical trial, the safety of subjects who participated in clinical trial and the clinical trial itself is objectively validated through the convocation and evaluation by Data Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurologic deficit of ≥ 4 points by NIHSS score
* Adults aged ≥19 years and ≤85 years. (Pre-stroke mRS must be 0 or 1; No significant pre-stroke disability)
* Subjects who can receive rtPA therapy within 4.5 hours after the onset of early symptoms of acute ischemic stroke.
* Subjects available for brain MRI (DWI, GRE/Susceptibility Weighted Imaging (SWI), FLAIR, MRA) scanning
* Subjects who consent to participate in this trial.

Exclusion Criteria:

* Patients with systemic allergic diseases or hypersensitivity to specific drugs.
* Patients who were diagnosed with myocardial infarction (MI) within the last 6 months.
* Patients who had arrhythmia causing clinical symptoms such as dyspnea or palpitation within the last 6 months.
* Patients showing the following abnormal ECG findings in stable condition at Emergency Room:

  * The range of pulse rate - under 55/min or exceed 120/min
  * 2nd or 3rd degree Atrioventricular (AV) block indicated in ECG
  * Congenital or acquired QT syndrome indicated in ECG
  * Pre-excitation syndrome indicated in ECG
* Patients with severe heart failure of New York Heart Association (NYHA) Class III or Class IV.
* Patients with fever (≥ 38℃) or infection signs which require antibiotic therapy at screening.
* Patients with pulmonary diseases (asthma, Chronic Obstruction Pulmonary disease, and active tuberculosis etc.) who have being recently been treated more than 1 month at screening.
* Patients with decreased hemoglobin (Hb< 10g/dL), decreased platelet count (PLT< 100,000/mm3) or hematocrit of <25% in complete blood count.
* Patients who have undergone hemodialysis and/or treatments due to nephropathies, acute or chronic renal failure at screening.
* Patients with a cancer in following conditions: diagnosed within 6 months before the screening time, or any treatment for cancer within the previous 6 months, or with recurrent/ metastatic cancer.
* Pregnant and lactating women. However, women of childbearing age can participate in the trial only when non-pregnancy is confirmed. Woman of childbearing age is defined as woman who is not definitely menopause and did not receive a surgical contraception.
* Patients who do not consent to use double barrier contraception during the trial period.
* Patients who have participated in other clinical trials of other drugs within the past 3 months. However, if they participated in observational studies and did not take drugs, they can participate in this trial.
* Patients who cannot participate in the trial according to the judgment of investigators.
* Those who cannot be administered with rtPA.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
The neurological improvement evaluated by the National Institute of Health Stroke Scale (NIHSS) | Change from 0 day at 28 days
  The neurological improvement evaluated by the National Institute of Health Stroke Scale (NIHSS) until 28 day in subjects with acute ischemic stroke requiring rtPA (recombinant tissue Plasminogen Activator) standard of care. The maximum total score is 42 points, which indicates the most critical condition and the minimum total score is 0, which indicates no neurologic deficit.

SECONDARY OUTCOMES:
Incidence of parenchymal hematoma observed on brain Computed Tomography (CT) scan | Day 1
  Incidence of parenchymal hematoma observed on brain Computed Tomography (CT) scan performed at 24±3 hours in accordance with European Cooperative Acute Stroke Study (ECASS) I and II criteria, after the administration of SP-8203 in conjunction with rtPA standard of care
The difference in the distribution of modified Rankin Scale (mRS) scores | Day 90
  The difference in the distribution of modified Rankin Scale (mRS) scores in subjects with acute ischemic stroke requiring rtPA standard of care. The 0-6 point-scales are scored according to symptoms with 0 point indicating no disability; the higher score denotes ofr the more severe degree of disability.
The change in the National Institute of Health Stroke Scale (NIHSS) scores | Change from 0 day at 90 days
  The change in the National Institute of Health Stroke Scale (NIHSS) scores until 90 day in subjects with acute ischemic stroke requiring rtPA standard of care. The maximum total score is 42 points, which indicates the most critical condition and the minimum total score is 0, which indicates no neurologic deficit.
The change in Barthel index | Change from 0 day at 90 days
  The change in Barthel index in subjects with acute ischemic stroke requiring rtPA standard of care
The fold change of infarct growth classified by modified Treatment in Cerebral Ischemia (mTICI) grade within 5 days | Day 5
  MRI (DWI) imaging outcomes
The number of occurrence and volume of intracranial hemorrhage classified by mTICI grade within 5 days | Day 5
  MRI (GRE) imaging outcomes
The incidence of serious adverse events | follow-up to 30 days after the last visit
  The incidence of serious adverse events
The rate of death | follow-up to 30 days after the last visit
  The rate of death due to any cause
The incidence rate of adverse events, and adverse drug reaction | follow-up to 30 days after the last visit
  The incidence rate of adverse events, and adverse drug reaction
The incidence of symptomatic Intracranial Hemorrhage (sICH) | within 5 days of administration
  The incidence of sICH occurring within 5 days of administration according to the definition described on the protocol
The Incidence of major systemic bleeding | within 5 days of administration
  The Incidence of major systemic bleeding according to the International Society of Thrombosis and Hemostasis (ISTH) definition

CONTACTS AND LOCATIONS:
Overall Officials: Jong Sung Kim, MD, Phd, Study Chair — Asan Medical Center; Dae-IL Chang, MD, Phd, Principal Investigator — Kyunghee University Medical Center; Kyung Mi Oh, MD, Phd, Principal Investigator — Korea University Guro Hospital; Jong-Ho Park, MD, Phd, Principal Investigator — Myongji Hospital; Kyung Bok Lee, MD, Phd, Principal Investigator — Soonchunhyang University Hospital; Sang Min Sung, MD, Phd, Principal Investigator — Pusan National University Hospital; Eung-Gyu Kim, MD, Phd, Principal Investigator — Inje University; Hee-Joon Bae, MD, Phd, Principal Investigator — Seoul National University Bundang Hospital; Jee-Hyun Kwon, MD, Phd, Principal Investigator — Ulsan University Hospital; Jae Gwan Cha, MD, Phd, Principal Investigator — Dong-A University Hospital; Man Seok Park, MD, Phd, Principal Investigator — Chonnam National University Hospital; Jong Moo Park, MD, Phd, Principal Investigator — Nowon Eulji Medical Center; Yang Ha Hwang, MD, Phd, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Asan Medical Center, Seoul, South Korea